CLINICAL TRIAL: NCT05205304
Title: The Role of Transdermal Carbon Dioxide in Malondialdehyde Level as Predictor of Ischemia Reperfusion Injury in Patients Underwent Abdominal Aortic Temporary Cross Clamp
Brief Title: The Role of Transdermal CO2 in MDA Level in Patient Underwent Abdominal Aortic Temporary Cross Clamp
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitas Airlangga (Other)
Responsible Party: Principal Investigator, Hari Daswin Pagehgiri, Resident of Thoracic, Cardiac, and Vascular Surgery Department, Universitas Airlangga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCVS UA
Record Dates: First submitted 2022-01-03; First posted 2022-01-25 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-01

CONDITIONS: Placenta Accreta
Keywords: Abdominal Aortic Cross Clamp
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Intervention Model Description: Subjects will be divided into two groups. The first group is treated with CO2 transdermal administration and the second group is the control group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment group (Experimental): Subjects will be treated with liquid carbon dioxide (D'oxyva) administered transdermally on the thumb after the Aortic Cross Clamp is removed
  Interventions: Drug: D'Oxyva
- Control group (No Intervention): Subject will not be treated with liquid carbon dioxide (D'oxyva)

INTERVENTIONS:
Drug: D'Oxyva — The transdermal CO2 was administered via non-invasive vaporization technique accommodated by deoxyhemoglobin vasodilator (D'Oxyva)
  Other Names: Transdermal CO2
  Arms: Treatment group

SUMMARY:
The Role of Transdermal Carbon Dioxide in Malondialdehyde Level as Predictor of Ischemia Reperfusion Injury in Patients Underwent Abdominal Aortic Temporary Cross Clamp

DETAILED DESCRIPTION:
Abdominal aortic temporary cross clamping procedures in patients with placenta accreta undergoing hysterectomy have been performed at Dr. Soetomo Hospital Surabaya for a period of 4 years. In the aortic cross-clamping procedure, an ischemic condition occurs, after the cross-clamp is released the distal tissue from the occlusion which was initially in an ischemic state gets blood flow suddenly (reperfusion) causing Ischemia Reperfusion Injury. This study aims to determine the effect of transdermal administration of carbon dioxide (CO2) as a protective factor for ischemia reperfusion injury in patients undergoing Abdominal Aorta Temporary Cross Clamp. The design of this study is experimental in patients who underwent Abdominal Aorta Temporary Cross Clamp. Subjects were divided into two groups. The first group was treated with CO2 transdermal administration and the second group was the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Placenta Accreta diagnosed with placental accreta index (PAI) based on the results of ultrasound and underwent Abdominal Aorta Clamping Surgery (Control of Bleeding in Accreta)

Exclusion Criteria:

* Patients with severe comorbid disorders based on previous clinical examination: chronic kidney disease, heart disease
* Patients with septic shock and sepsis
* Patients with peripheral artery disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Malondyaldehyde | Basal, 1 hour after aortic cross clamp off
  The malondyaldehyde concentration of the patient's serum measured by ELISA test method

CONTACTS AND LOCATIONS:
Locations (1):
- Hari Daswin Pagehgiri, Surabaya, Bali, Indonesia